CLINICAL TRIAL: NCT03710421
Title: Phase I Study to Evaluate Cellular Immunotherapy Using Memory-Enriched T Cells Lentivirally Transduced to Express a CS1-Targeting, Hinge-Optimized, 41BB-Costimulatory Chimeric Antigen Receptor and a Truncated EGFR Following Lymphodepleting Chemotherapy in Adult Patients With CS1+ Multiple Myeloma
Brief Title: CS1-CAR T Therapy Following Chemotherapy in Treating Patients With Relapsed or Refractory CS1 Positive Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17403; NCI-2018-02022 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17403 (Other: City of Hope Medical Center)
Record Dates: First submitted 2018-10-05; First posted 2018-10-18 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; fludarabine; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (leukapheresis, chemotherapy, CS-1 CAR T therapy) (Experimental): Patients undergo leukapheresis over 2-4 hours. Beginning 3-4 weeks, patients receive cyclophosphamide IV on days -4 and/or -3 or fludarabine IV and cyclophosphamide IV on days -5 to -3. Patients then undergo CS1-CAR T therapy over 10-15 minutes on day 0.
  Interventions: Procedure: CS1-CAR T Therapy; Drug: Cyclophosphamide; Drug: Fludarabine; Procedure: Leukapheresis

INTERVENTIONS:
Procedure: CS1-CAR T Therapy — Undergo CS1-CAR T therapy
  Other Names: CS1-CAR T Infusion; CS1-CAR T-cell Therapy
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis

SUMMARY:
This phase I trial studies the side effects and best dose of CS1-chimeric antigen receptor (CAR) T therapy after chemotherapy in treating patients who have CS1 positive multiple myeloma that has come back (relapsed) or does not respond to treatment (refractory). Immune cells can be engineered to kill multiple myeloma cells by inserting a piece of deoxyribonucleic acid (DNA) into the immune cells using a lentiviral vector such as CS1, that allows them to recognize multiple myeloma cells. These engineered immune cells, CS1-CAR T cells, may kill multiple myeloma cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and tolerability of intravenous (i.v.) delivered autologous CS1-CAR T cells for research participants with CS1+ recurrent/refractory multiple myeloma (MM).

SECONDARY OBJECTIVES:

I. Evaluate the response rates at days 28, 100, and 180 post CAR T cell infusion.

II. Measure the persistence of CS1-CAR T cells in blood and marrow. III. Measure phenotype and anti-tumor functionality of CS1-CAR T cells in marrow and blood.

IV. Measure the levels of cytokines in blood and marrow, and soluble CS-1 in blood post infusion as a surrogate indicator of CAR T cell activity.

V. Evaluate CS-1 expression on MM cancer cells before, during and at progressive disease (PD) to determine antigenic loss.

EXPLORATORY OBJECTIVE:

I. Describe the percentage of MM cells that express CS-1 surface marker before, during and at PD.

OUTLINE: This is a dose-escalation study of CS1-CAR T cells.

Patients undergo leukapheresis over 2-4 hours. Beginning 3-4 weeks, patients receive cyclophosphamide intravenously (IV) on days -4 and/or -3 or fludarabine IV and cyclophosphamide IV on days -5 to -3. Patients then undergo CS1-CAR T therapy over 10-15 minutes on day 0.

After completion of study treatment, patients are followed up at 1 day, at least every 2 days for up to a minimum of 14 days, weekly for 1 month, monthly for 1 year, then periodically for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines.
* Karnofsky Performance Status (KPS) of >= 70%.
* Life expectancy >= 16 weeks.
* Participant must have a confirmed diagnosis of active MM as defined by the International Myeloma Working Group (IMWG) criteria.
* Participant must have a confirmed CS1+ MM as evaluated by City of Hope (COH) Pathology Core.
* Participant must have measurable disease defined as meeting at least one of the criteria below:

  * Serum M-protein >= 0.5 g/dL.
  * Urine M-protein >= 200 mg/24 hour.
  * Involved serum free light chain (sFLC) level >= 10 mg/dL with abnormal kappa/lambda ratio.
  * Measurable biopsy-proven plasmacytomas (>= 1 lesion that has a single diameter >= 2 cm)
  * Bone marrow plasma cells >= 30%.
* Participant must have relapsed or refractory disease after all 3 prior treatment regimens with the following requirements:

  * Participant must have received prior treatment with an immunomodulatory agent.
  * Participant must have received prior treatment with a proteasome inhibitor.
  * Participant must have received prior treatment with an anti-CD38 antibody.
  * Participants must be refractory to last line of therapy prior to study enrollment (refractory myeloma is defined as disease that is nonresponsive, progression on treatment, or shows progression within 60 days after the last prior line of therapy).
  * Participants who were not candidates to receive one or more of the above treatments are eligible; however, the reason must be clearly documented in the case report form.
  * Note: induction chemotherapy, autologous stem-cell transplantation (ASCT), and maintenance therapy should be considered as 1 "regimen."
* Additionally, if a participation underwent autologous transplant he/she be >= 90 days from transplant at the time of enrollment.
* Total serum bilirubin =< 2.0 mg/dL.
* Participants with Gilbert syndrome may be included if their total bilirubin is =< 3.0.
* Aspartate aminotransferase (AST) < 2.5 x upper limit of normal (ULN).
* Alanine aminotransferase (ALT) < 2.5 x ULN.
* Serum creatinine =< 2.5 x ULN or estimated creatinine clearance of >= 40 mL/min per the Cockcroft-Gault formula, and the participant is not on hemodialysis.
* Absolute neutrophil count >= 1000/uL. Transfusions and growth factors must not be used to meet these requirements at initial screening.
* Hemoglobin (Hb) >= 8 g/dl. Transfusions and growth factors must not be used to meet these requirements at initial screening.
* Platelet count >= 50,000/uL (>= 30,000/uL if bone marrow plasma cells are >= 50% of cellularity). Transfusions and growth factors must not be used to meet these requirements at initial screening.
* Left ventricular ejection fraction >= 45% within 8 weeks before enrollment.
* Oxygen (O2) saturation >= 92%.
* Women of childbearing potential (WOCBP): Negative urine or serum pregnancy test.
* If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only).

Exclusion Criteria:

* Prior allogeneic stem cell transplantation.
* Autologous transplantation =< 90 days of enrollment.
* Growth factors within 14 days of enrollment.
* Platelet transfusions within 7 days of enrollment.
* Epstein-Barr virus (EBV) positivity by polymerase chain reaction (PCR) at the time of enrollment
* Participants receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy.
* Participants with known additional malignancy that is progressing or required active treatment within the last 2 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Participants with toxicities from prior therapies, with the exception of peripheral neuropathy attributable to bortezomib, that have not recovered to grade =< 2 according to the Common Terminology Criteria for Adverse Events (CTCAE) 5.0 criteria or to the subject's prior baseline.
* Participants with known active hepatitis B or C infection; research participants who are human immunodeficiency virus (HIV) positive based on testing performed within 4 weeks of enrollment; research participants with any signs or symptoms of active infection, positive blood cultures or radiological evidence of infections.
* Participants with active auto-immune disease, including connective tissue disease, sarcoidosis, multiple sclerosis, inflammatory bowel disease or have a history of severe (as judged by the principal investigator) autoimmune disease that will require prolonged immunosuppressive therapy.
* Have New York Heart Association (NYHA) Class III or IV heart failure, unstable angina, or a history of recent (within 6 months) myocardial infarction.
* Participants with a history or presence of clinically relevant central nervous system (CNS) pathology such as uncontrolled seizure disorder, stroke, severe brain injuries, dementia, cerebellar disease or psychosis.
* Participants with known active central nervous system (CNS) involvement by malignancy. Subjects with prior CNS disease that has been effectively treated will be eligible if treatment was completed at least 3 months prior to enrollment with no evidence of symptomatic disease and stable abnormalities on repeat imaging.
* Participants with plasma cell leukemia (PCL) or symptomatic amyloidosis. However, participants with a prior history of PCL are not excluded.
* Participants with any known contraindications to leukapheresis, cyclophosphamide, fludarabine, cetuximab or tocilizumab.
* Dependence on corticosteroids.

  * Defined as doses of corticosteroids of greater than or equal to 10 mg/day of prednisone or equivalent doses of other corticosteroids.
  * Note: Topical and inhaled corticosteroids in standard doses and physiologic replacement for subjects with adrenal insufficiency are allowed.
* Participants with inadequate venous access for leukapheresis, and who are either unable to or unwilling to have a supportive line (temporary or other) placed for the procedure.
* Females only: Pregnant or breastfeeding.
* Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns with clinical study procedures.
* Prospective subjects who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-23 (Actual); Primary Completion 2026-03-24 (Estimated); Study Completion 2026-03-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) and all other toxicities | Up to 12 months
  Tables will be created to summarize all toxicities and side effects by organ, severity (Common Terminology Criteria for Adverse Events version 5.0), and attribution. Rates and associated 90% confidence limits will be estimated for participants experiencing DLTs.
Incidence of all other toxicities | Up to 15 years
  Will be assessed by Common Terminology Criteria for Adverse Events version 5.0. Will include cytokine release syndrome (CRS) based on the revised CRS grading system, and heart failure based on New York Heart Association criteria.
Opportunistic infections | Up to 15 years
Prolonged lymphopenia (lasting more than 12 weeks) | Up to 15 years

SECONDARY OUTCOMES:
Disease response | Up to 180 days
  Disease status will be evaluated based on the International Myeloma Working Group for Multiple Myeloma. Descriptive statistics will be provided for patient demographics, phenotype and functionality of modified T cells as well as anti-tumor immune response.
Expansion/persistence of chimeric antigen receptor (CAR) T cells | At 28 days post CAR T cell infusion
  Rates and associated 90% confidence limits will be estimated for participants achieving persistence/expansion of T cells at 28 days. To further study T cell expansion and persistence, area under the curve of log10 copies/ug of genomic deoxyribonucelic acid over the 28 day period post T cell infusion will be calculated for each participant and presented both graphically and using descriptive statistics.
Phenotype and anti-tumor functionality of modified T cells in marrow and blood | Up to 15 years
  Descriptive statistics will be provided for patient demographics, phenotype and functionality of modified T cells as well as anti-tumor immune response.
Cytokine and soluble CS-1 levels in blood and marrow | Up to 15 years
  Statistical and graphical methods will be used to describe the cytokine levels (marrow and blood) over the study period.
Disease free survival (DFS) | At 12 months
  Rates and associated 90% confidence limits will be estimated for participants experiencing DFS. Kaplan Meier methods will be used to describe the survival distributions both statistically and graphically.
Progression-free survival | At 12 months
  Kaplan Meier methods will be used to describe the survival distributions both statistically and graphically.
CS1 expression on multiple myeloma cells | Baseline up to 15 years

OTHER OUTCOMES:
MM cells that are CS-1 positive | Up to 15 years
  Descriptive statistics are provided for the percentage of MM cells that express CS-1 surface marker.

CONTACTS AND LOCATIONS:
Overall Officials: Myo Htut, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States